CLINICAL TRIAL: NCT00040547
Title: Safety and Tolerability Study of Farnesyl Protein Transferase Inhibitor (FPTI) in Combination With Docetaxel in Advanced Solid Tumors
Brief Title: Farnesyl Protein Transferase Inhibitor (FPTI) in Combination With Docetaxel in Advanced Solid Tumors (Study P01964)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01964
Record Dates: First submitted 2002-06-28; First posted 2002-07-01 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Neoplasms
Keywords: Cancer-Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — 2-(2-oxo-2-((3,7,11-trimethyl-2,6,10-dodecatrienyl)oxy)aminoethyl)phosphonic acid, (2,2-dimethyl-1-oxopropoxy)methyl ester sodium

INTERVENTIONS:
Drug: Farnesyl Protein Transferase Inhibitor

SUMMARY:
The purpose of this study is to determine the safety and tolerability of an oral Farnesyl Protein Transferase Inhibitor (SCH 66336) when given in combination with intravenous docetaxel in cancer patients with advanced solid tumors.

ELIGIBILITY:
Inclusion:

* Male or Female
* Measurable or evaluable disease
* No more than 2 prior chemotherapy regimens.
* Age greater than or equal to 18.
* Karnofsky Performance Status greater than or equal to 70%.
* Meets protocol requirements for specified laboratory values.
* No manifestations of a malabsorption syndrome.
* Written informed consent and cooperation of patient
* Appropriate use of effective contraception if of child-bearing potential.

Exclusion:

* Acute or chronic leukemia or multiple myeloma.
* Evidence of 2 or more active malignancies, expect for in situ or adequately treated basal or squamous cell skin cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2001-06; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events
Laboratory Tests
ECG

SECONDARY OUTCOMES:
Physical Exam
Pharmacokinetics
Tumor Response